CLINICAL TRIAL: NCT07167264
Title: Evaluation of a Combined PGHD-AI Intelligent Model for the Nutritional Assessment and Intervention of Patients After Radical Surgery for Pancreatic Cancer.
Brief Title: PGHD-AI Intelligent Model for the Nutritional Assessment and Intervention of Patients After Radical Surgery for Pancreatic Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Long, Head of pancreatic surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PGHD-2025
Record Dates: First submitted 2025-09-02; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients use the APP to check in daily and record PGHD data, combined with offline routine follow-up, nutritional assessment and intervention.
  Interventions: Other: PGHD's AI intelligent model(APP)
- Control group (No Intervention): Patients received routine outpatient follow-up and nutritional assessment by investigator.

INTERVENTIONS:
Other: PGHD's AI intelligent model(APP) — To collect patient PRO (physical strength, pain, defecation, appetite, weight, etc.) data through the PGHD's AI intelligent model(APP), and use corpus collection cards, facial photography and other technologies to collect PGHD characteristic phenotypes.
  Arms: Intervention group

SUMMARY:
This study will collect patient PRO (physical strength, pain, defecation, appetite, weight, etc.) data through the APP, use corpus collection cards, facial photography and other technologies to collect PGHD characteristic phenotypes, and then combine artificial intelligence technology to train and cultivate agents (agents) to carry out joint offline routine follow-up of patients after radical pancreatic cancer resection to evaluate the feasibility of nutritional risk assessment intervention. Thus, the feasibility of artificial intelligence prediction of health status is verified, and an efficient follow-up tool and nutritional support evaluation plan are provided for the management of pancreatic cancer patients throughout the course of the disease, so as to improve the treatment prognosis and quality of life of pancreatic cancer patients.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled exploratory clinical trial to recruit 200 patients after radical pancreatic cancer resection.

Screening eligible subjects will be randomly assigned to the test group and the control group, and the randomization stratification factors include: age, gender, TNM stage, ECOG score, baseline BMI.

The experimental group and the control group received offline routine follow-up combined with PGHD-AI's APP management and routine outpatient follow-up, respectively, to compare the prediction of nutritional status risk and intervention response.

The study period is 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, and voluntarily signed the informed consent form to participate in the study;
2. Meet the clinical and pathological diagnostic criteria for pancreatic cancer (ICD-10:C25);
3. After radical surgery, fully recovered from surgery at randomization;
4. ECOG PS score 0-1 ;
5. Have objective conditions to complete follow-up and examination during the study process.

Exclusion Criteria:

1. Patients or their families are willing to use the APP;
2. Current history or past history of metastatic or locally recurrent pancreatic cancer;
3. Combined with other serious organ dysfunctions (such as severe liver and kidney insufficiency, heart failure, etc.);
4. Women who are currently pregnant or lactating;
5. History of other tumor diseases in the past;
6. Other conditions that the study deems unsuitable for participation in the study, including but not limited to: patients with serious or uncontrollable medical conditions, safety risks, interference with the interpretation of study results, and impact on study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and/or improvement rate | 12 months after enrollment
The progression free survival | 12 months after enrollment
The overall survival time | 12 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China